CLINICAL TRIAL: NCT00193713
Title: A Randomized, Double-Blind, Olanzapine-Referenced, Parallel-Group Safety and Efficacy Study of Flexible Doses of Bifeprunox in the Long-term Treatment of Schizpohrenia (Extension of S1543003)
Brief Title: Bifeprunox in the Treatment of Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S154.3.004
Record Dates: First submitted 2005-09-11; First posted 2005-09-19 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2007-01

CONDITIONS: Schizophrenia
Keywords: double-blind study in the treatment of schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — bifeprunox

INTERVENTIONS:
Drug: bifeprunox

SUMMARY:
Study of the long-term efficacy and safety of bifeprunox in the treatment of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of schizophrenia
* understand nature of study
* able to be managed in out-patient setting for long-term bifeprunox treatment

Exclusion Criteria:

* current primary diagnosis other than schizophrenia
* suicide risk
* diagnosis or history of substance abuse
* uncontrolled hypertension

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-05; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals